CLINICAL TRIAL: NCT02976038
Title: A Multicenter, Open-Label Phase 2 Extension Trial to Characterize the Long-term Safety and Tolerability of Subcutaneous Elamipretide in Subjects With Genetically Confirmed Primary Mitochondrial Myopathy (PMM)
Brief Title: Open-Label Extension Trial to Characterize the Long-term Safety and Tolerability of Elamipretide in Subjects With Genetically Confirmed Primary Mitochondrial Myopathy (PMM)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Registration trial did not meet the primary end points
Sponsor: Stealth BioTherapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPIMM-203
Record Dates: First submitted 2016-11-18; First posted 2016-11-29 (Estimated); Results first posted 2021-12-17 (Actual); Last update posted 2021-12-17 (Actual); Status verified 2021-11

CONDITIONS: Primary Mitochondrial Disease
Keywords: Primary Mitochondrial Disease; Stealth; elamipretide
MeSH Terms: interventions — arginyl-2,'6'-dimethyltyrosyl-lysyl-phenylalaninamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- elamipretide (Experimental): Open-label once daily subcutaneous injection of 40mg elamipretide
  Interventions: Drug: elamipretide

INTERVENTIONS:
Drug: elamipretide — 40 mg, subcutaneous injections (in the abdomen) daily for the shortest of the following: 260 weeks; regulatory approval and commercial availability of elamipretide in the subject's respective country; or termination of the clinical development for elamipretide in subjects with PMD.

SUMMARY:
This is a Phase 2 Open-Label extension study to evaluate the long term safety and tolerability of daily elamipretide injections in patients with genetically confirmed Primary Mitochondrial Disease who previously participated in the SPIMM-202 Clinical Trial

DETAILED DESCRIPTION:
This open-label, non-comparative, extension trial will enroll subjects with genetically confirmed PMD who have completed the End-of-Study Visit in the SPIMM-202 trial. Subjects who do not discontinue or withdraw from the trial will receive treatment with 40 mg SC elamipretide for the shortest of the following: 260 weeks; regulatory approval and commercial availability of elamipretide in the subject's respective country; or termination of the clinical development for elamipretide in subjects with PMD.

ELIGIBILITY:
Inclusion Criteria:

* Investigator determines the subject can, and subject agrees to, adhere to the trial requirements for the length of the trial including self-administration (by subject or trained caregiver) of the study drug
* Subject completed the End-of-Study Visit in SPIMM-202

Exclusion Criteria:

* Subject has any prior or current medical condition that, in the judgment of the Investigator, would prevent the subject from safely participating in and/or completing all trial requirements
* Subject has received any investigational compound (excluding elamipretide) and/or has participated in another interventional clinical trial within 30 days prior to the SPIMM-203 Baseline Visit (excluding SPIMM-202) or is concurrently enrolled in any non-interventional research of any type judged to be scientifically or medically incompatible with the trial as deemed by the Investigator in consultation with the Sponsor
* Subject experienced an adverse reaction attributed to study drug resulting in permanent discontinuation of study drug in the SPIMM-202 trial.
* Female subjects who are pregnant, planning to become pregnant, or lactating
* Subject has undergone an in-patient hospitalization within the 1 month prior to the SPIMM-203 Baseline Visit

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2020-03-09 (Actual); Study Completion 2020-04-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jim Carr, PharmD, Study Director — Stealth BioTherapeutics
Locations (4):
- United States (4):
  - University of California, San Diego, California
  - Massachusetts General Hospital, Boston, Massachusetts
  - Akron Children's Hospital, Akron, Ohio
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Elamipretide
Started | 28
Completed | 0
Not Completed | 28
Not completed — Physician Decision | 22
Not completed — Withdrawal by Subject | 3
Not completed — Lost to Follow-up | 2
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Population: All participants for whom Baseline measurements were taken.
Arm/Group | Elamipretide
Number analyzed (Participants) | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.8 (11.30)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 27
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 27
  More than one race | 1
  Unknown or Not Reported | 0
Baseline weight [Mean (Standard Deviation); unit: kg] | 65.93 (14.614)

OUTCOME MEASURES:

1. Primary Outcome: Distance Walked on Six Minute Walk Test
Description: Change From Baseline in Distance Walked (meters) on the Six-Minute Walk Test by Visit
Time Frame: Baseline, Month 3, Month 6 and Every 26 weeks for up to 160 weeks
Population: All participants for whom Change From Baseline in Distance Walked (meters) on the Six-Minute Walk Test by Visit was measured.
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Elamipretide
Number analyzed (Participants) | 28
meters
  Week 13 | 3.6 (52.68)
  Week 26: number analyzed (Participants) | 27
  Week 26 | -8.6 (56.33)
  Week 52: number analyzed (Participants) | 25
  Week 52 | -17.6 (70.60)
  Week 78: number analyzed (Participants) | 24
  Week 78 | -26.2 (73.17)
  Week 104: number analyzed (Participants) | 22
  Week 104 | -20.9 (77.78)
  Week 130: number analyzed (Participants) | 20
  Week 130 | -18.9 (76.94)
  Week 156: number analyzed (Participants) | 1
  Week 156 | -35.0 (NA) — Only 1 participant.
  End of Trial (Week 160): number analyzed (Participants) | 19
  End of Trial (Week 160) | -54.0 (70.30)

2. Secondary Outcome: EuroQol 5 Dimensions 5 Levels (EQ-5D-5L)
Description: EuroQol 5 dimensions 5 levels (EQ-5D-5L) by visit. Count of participants per arm, or severity level of dimension. Measures 5 dimensions: mobility, self-care, usual activities, pain/discomfort, anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. Score ranges from 5-25 with lower score=better outcome, and higher score means a worse outcome.
Time Frame: Baseline, Month 3, Month 6 and Every 26 weeks for up to 160 weeks
Population: All participants for whom EQ-5D-5L was measured. Trial was terminated early.
Measure: Count of Participants; unit: Participants
Groups:
- No Problem: Participant reports symptom is "no problem"
- Slight Problem: Participant reports symptom is a "slight problem"
- Moderate Problem: Participant reports symptom is a "moderate problem"
- Severe Problem: Participant reports symptom is a "severe problem"
- Extreme Problem: Participant reports symptom is an "extreme problem"
Arm/Group | No Problem | Slight Problem | Moderate Problem | Severe Problem | Extreme Problem
Number analyzed (Participants) | 28 | 28 | 28 | 28 | 28
Participants
  Baseline: Anxiety/Depression | 12 | 8 | 4 | 3 | 1
  Baseline: : Mobility | 2 | 10 | 11 | 5 | 0
  Baseline: : Pain/Discomfort | 4 | 5 | 15 | 4 | 0
  Baseline: : Self-Care | 12 | 10 | 5 | 0 | 1
  Baseline: : Usual Activities | 5 | 7 | 12 | 4 | 0
  Week 13 Anxiety/Depression | 16 | 6 | 5 | 1 | 0
  Week 13 : Mobility | 7 | 7 | 12 | 1 | 1
  Week 13 : Pain/Discomfort | 4 | 12 | 8 | 3 | 1
  Week 13 : Self-Care | 18 | 7 | 2 | 0 | 1
  Week 13 : Usual Activities | 6 | 15 | 5 | 0 | 2
  Week 26 Anxiety/Depression: number analyzed (Participants) | 27 | 27 | 27 | 27 | 27
  Week 26 Anxiety/Depression | 16 | 6 | 5 | 0 | 0
  Week 26 : Mobility: number analyzed (Participants) | 27 | 27 | 27 | 27 | 27
  Week 26 : Mobility | 5 | 6 | 12 | 4 | 0
  Week 26 : Pain/Discomfort: number analyzed (Participants) | 27 | 27 | 27 | 27 | 27
  Week 26 : Pain/Discomfort | 8 | 11 | 5 | 2 | 1
  Week 26 : Self-Care: number analyzed (Participants) | 27 | 27 | 27 | 27 | 27
  Week 26 : Self-Care | 17 | 7 | 3 | 0 | 0
  Week 26 : Usual Activities: number analyzed (Participants) | 27 | 27 | 27 | 27 | 27
  Week 26 : Usual Activities | 6 | 13 | 7 | 1 | 0
  Week 56 Anxiety/Depression: number analyzed (Participants) | 25 | 25 | 25 | 25 | 25
  Week 56 Anxiety/Depression | 14 | 5 | 4 | 1 | 1
  Week 56 : Mobility: number analyzed (Participants) | 25 | 25 | 25 | 25 | 25
  Week 56 : Mobility | 6 | 6 | 4 | 9 | 0
  Week 56 : Pain/Discomfort: number analyzed (Participants) | 25 | 25 | 25 | 25 | 25
  Week 56 : Pain/Discomfort | 6 | 8 | 9 | 2 | 0
  Week 56 : Self-Care: number analyzed (Participants) | 25 | 25 | 25 | 25 | 25
  Week 56 : Self-Care | 16 | 6 | 2 | 1 | 0
  Week 56: Usual Activities: number analyzed (Participants) | 25 | 25 | 25 | 25 | 25
  Week 56: Usual Activities | 8 | 9 | 5 | 3 | 0
  Week 78 Anxiety/Depression: number analyzed (Participants) | 24 | 24 | 24 | 24 | 24
  Week 78 Anxiety/Depression | 12 | 6 | 3 | 2 | 1
  Week 78 : Mobility: number analyzed (Participants) | 24 | 24 | 24 | 24 | 24
  Week 78 : Mobility | 5 | 8 | 8 | 2 | 1
  Week 78 : Pain/Discomfort: number analyzed (Participants) | 24 | 24 | 24 | 24 | 24
  Week 78 : Pain/Discomfort | 4 | 14 | 5 | 1 | 0
  Week 78 : Self-Care: number analyzed (Participants) | 24 | 24 | 24 | 24 | 24
  Week 78 : Self-Care | 15 | 6 | 2 | 1 | 0
  Week 78 : Usual Activities: number analyzed (Participants) | 24 | 24 | 24 | 24 | 24
  Week 78 : Usual Activities | 5 | 12 | 6 | 1 | 0
  Week 104 Anxiety/Depression: number analyzed (Participants) | 22 | 22 | 22 | 22 | 22
  Week 104 Anxiety/Depression | 10 | 7 | 4 | 0 | 1
  Week 104 : Mobility: number analyzed (Participants) | 22 | 22 | 22 | 22 | 22
  Week 104 : Mobility | 4 | 5 | 10 | 2 | 1
  Week 104 : Pain/Discomfort: number analyzed (Participants) | 22 | 22 | 22 | 22 | 22
  Week 104 : Pain/Discomfort | 5 | 8 | 9 | 0 | 0
  Week 104 : Self-Care: number analyzed (Participants) | 22 | 22 | 22 | 22 | 22
  Week 104 : Self-Care | 15 | 4 | 1 | 2 | 0
  Week 104 : Usual Activities: number analyzed (Participants) | 22 | 22 | 22 | 22 | 22
  Week 104 : Usual Activities | 3 | 13 | 4 | 2 | 0
  Week 130 Anxiety/Depression: number analyzed (Participants) | 22 | 22 | 22 | 22 | 22
  Week 130 Anxiety/Depression | 7 | 8 | 3 | 4 | 0
  Week 130 : Mobility: number analyzed (Participants) | 22 | 22 | 22 | 22 | 22
  Week 130 : Mobility | 7 | 4 | 8 | 3 | 0
  Week 130 : Pain/Discomfort: number analyzed (Participants) | 22 | 22 | 22 | 22 | 22
  Week 130 : Pain/Discomfort | 7 | 6 | 5 | 4 | 0
  Week 130 : Self-Care: number analyzed (Participants) | 22 | 22 | 22 | 22 | 22
  Week 130 : Self-Care | 14 | 5 | 1 | 2 | 0
  Week 130 : Usual Activities: number analyzed (Participants) | 22 | 22 | 22 | 22 | 22
  Week 130 : Usual Activities | 6 | 8 | 6 | 1 | 1
  Week 156 Anxiety/Depression: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1
  Week 156 Anxiety/Depression | 0 | 0 | 1 | 0 | 0
  Week 156 : Mobility: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1
  Week 156 : Mobility | 1 | 0 | 0 | 0 | 0
  Week 156 : Pain/Discomfort: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1
  Week 156 : Pain/Discomfort | 0 | 0 | 1 | 0 | 0
  Week 156 : Self-Care: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1
  Week 156 : Self-Care | 1 | 0 | 0 | 0 | 0
  Week 156 : Usual Activities: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1
  Week 156 : Usual Activities | 0 | 1 | 0 | 0 | 0
  End of Study (Week 160) Anxiety/Depression: number analyzed (Participants) | 21 | 21 | 21 | 21 | 21
  End of Study (Week 160) Anxiety/Depression | 9 | 6 | 4 | 1 | 1
  End of Study (Week 160) : Mobility: number analyzed (Participants) | 21 | 21 | 21 | 21 | 21
  End of Study (Week 160) : Mobility | 3 | 5 | 9 | 4 | 0
  21End of Study (Week 160) : Pain/Discomfort: number analyzed (Participants) | 21 | 21 | 21 | 21 | 21
  21End of Study (Week 160) : Pain/Discomfort | 4 | 7 | 8 | 2 | 0
  End of Study (Week 160) : Self-Care: number analyzed (Participants) | 21 | 21 | 21 | 21 | 21
  End of Study (Week 160) : Self-Care | 9 | 8 | 3 | 1 | 0
  End of Study (Week 160) : Usual Activities: number analyzed (Participants) | 21 | 21 | 21 | 21 | 21
  End of Study (Week 160) : Usual Activities | 5 | 7 | 6 | 2 | 1

3. Secondary Outcome: Euroquol Visual Analog Scale
Description: Euroquol Visual Analog Scale (EQ VAS): A patient-reported measure. The visual scale is numbered from 0 to 100, participants are directed as follows:
  "100 means the best health you can imagine, 0 means the worst health you can imagine. Mark an X on the scale to indicate how your health is TODAY." Higher scores mean better outcome, lower scores mean worse outcome.
Time Frame: Baseline, Month 3, Month 6 and Every 26 weeks for up to 160 weeks
Population: All participants for whom EQ VAS was measured. Trial was terminated early.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Elamipretide
Number analyzed (Participants) | 28
score on a scale
  Baseline | 65.29 (17.83)
  Week 13: number analyzed (Participants) | 27
  Week 13 | 65.44 (22.68)
  Week 26: number analyzed (Participants) | 27
  Week 26 | 62.70 (21.23)
  Week 52: number analyzed (Participants) | 27
  Week 52 | 70.52 (21.27)
  Week 78: number analyzed (Participants) | 24
  Week 78 | 64.88 (22.18)
  Week 104: number analyzed (Participants) | 22
  Week 104 | 67.23 (21.75)
  Week 130: number analyzed (Participants) | 22
  Week 130 | 72.18 (21.38)
  Week 156: number analyzed (Participants) | 1
  Week 156 | 60.00 (NA) — Only 1 participant, so there is no standard deviation
  End of Trial (Week 160): number analyzed (Participants) | 21
  End of Trial (Week 160) | 60.48 (23.28)

4. Secondary Outcome: NeuroQOL Fatigue Questionnaire
Description: Change from baseline in NeuroQOL Fatigue Questionnaire by visit. Questionnaire is comprised of 8 questions measuring participants incidence of fatigue affecting activities of daily living. Participants respond by choosing one of the following: 1=never, 2=rarely, 3=sometimes, 4=often, 5=always, with a lower score meaning a better outcome with fatigue affecting participant less, and high score meaning a worse outcome, with fatigue affecting the participant more. Total raw scores range from 8-40. Scores were converted to percentages: range0-100%. Change from baseline score: negative number means improved from baseline, positive number means worsened compared to baseline.
Time Frame: Baseline, Month 3, Month 6 and Every 26 weeks for up to 160 weeks
Population: All participants for whom Neuro-Qol Fatigue was measured. Trial was terminated early.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Elamipretide
Number analyzed (Participants) | 28
score on a scale
  Week 13 | -8.39 (16.43)
  Week 26: number analyzed (Participants) | 27
  Week 26 | -9.33 (16.40)
  Week 52: number analyzed (Participants) | 25
  Week 52 | -10.88 (17.48)
  Week 78: number analyzed (Participants) | 24
  Week 78 | -6.79 (17.07)
  Week 104: number analyzed (Participants) | 22
  Week 104 | -8.27 (18.61)
  Week 130: number analyzed (Participants) | 22
  Week 130 | -6.77 (15.69)
  Week 156: number analyzed (Participants) | 1
  Week 156 | 13.00 (NA) — Only 1 participant was measured.
  End of Study (Week 21 up to Week 160): number analyzed (Participants) | 21
  End of Study (Week 21 up to Week 160) | -2.67 (17.38)

5. Secondary Outcome: Patient Global Assessment : Categorical
Description: Patient Global Assessment [PGA] Score by Visit, count of participants. Patient-reported current health status by visit. PGA Scale is as follows: 1=Excellent, 2=Very good, 3=Good, 4=Fair, and 5=Poor. Total score ranges from 1-5. Higher score means worse health status, means worse outcome.
Time Frame: Baseline, Month 3, Month 6 and Every 26 weeks for up to 160 weeks
Population: All participants for whom PGA was measured. Trial was terminated early.
Measure: Count of Participants; unit: Participants
Arm/Group | Elamipretide
Number analyzed (Participants) | 28
Participants
  Baseline: Excellent | 1
  Baseline: Fair | 11
  Baseline: Good | 9
  Baseline: Poor | 5
  Baseline: Very Good | 2
  Week 13: number analyzed (Participants) | 26
  Week 13: Excellent | 0
  Week 13: Fair | 6
  Week 13: Good | 12
  Week 13: Poor | 2
  Week 13: Very Good | 6
  Week 26: number analyzed (Participants) | 27
  Week 26: Excellent | 1
  Week 26: Fair | 10
  Week 26: Good | 8
  Week 26: Poor | 3
  Week 26: Very Good | 5
  Week 52: number analyzed (Participants) | 25
  Week 52: Excellent | 0
  Week 52: Fair | 3
  Week 52: Good | 13
  Week 52: Poor | 4
  Week 52: Very Good | 5
  Week 78: number analyzed (Participants) | 24
  Week 78: Excellent | 0
  Week 78: Fair | 7
  Week 78: Good | 10
  Week 78: Poor | 4
  Week 78: Very Good | 3
  Week 104: number analyzed (Participants) | 22
  Week 104: Excellent | 0
  Week 104: Fair | 7
  Week 104: Good | 8
  Week 104: Poor | 2
  Week 104: Very Good | 5
  Week 130: number analyzed (Participants) | 22
  Week 130: Excellent | 1
  Week 130: Fair | 6
  Week 130: Good | 10
  Week 130: Poor | 4
  Week 130: Very Good | 1
  Week 156: number analyzed (Participants) | 1
  Week 156: Excellent | 0
  Week 156: Fair | 1
  Week 156: Good | 0
  Week 156: Poor | 0
  Week 156: Very Good | 0
  End of Study End of Study (Week 21 up to Week 160): number analyzed (Participants) | 21
  End of Study End of Study (Week 21 up to Week 160): Excellent | 0
  End of Study End of Study (Week 21 up to Week 160): Fair | 8
  End of Study End of Study (Week 21 up to Week 160): Good | 9
  End of Study End of Study (Week 21 up to Week 160): Poor | 3
  End of Study End of Study (Week 21 up to Week 160): Very Good | 1

6. Secondary Outcome: Patient Global Assessment: Continuous Variable
Description: Patient Global Assessment [PGA] Score by Visit, Patient-reported current health status by visit. PGA Scale is as follows: 1=Excellent, 2=Very good, 3=Good, 4=Fair, and 5=Poor. Total score ranges from 1-5. Higher score means worse health status, lower score means worse outcome.
Time Frame: Baseline, Month 3, Month 6 and Every 26 weeks for up to 160 weeks
Population: All participants for whom Change From Baseline in Patient Global Assessment was measured.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Elamipretide
Number analyzed (Participants) | 28
score on a scale
  Baseline | 3.61 (0.99)
  Week 13: number analyzed (Participants) | 26
  Week 13 | 3.15 (0.88)
  Week 26: number analyzed (Participants) | 27
  Week 26 | 3.15 (0.88)
  Week 52: number analyzed (Participants) | 25
  Week 52 | 3.24 (0.97)
  Week 78: number analyzed (Participants) | 24
  Week 78 | 3.50 (0.93)
  Week 104: number analyzed (Participants) | 22
  Week 104 | 3.27 (0.94)
  Week 130: number analyzed (Participants) | 22
  Week 130 | 3.50 (1.01)
  Week 156: number analyzed (Participants) | 1
  Week 156 | 4.00 (NA) — Only 1 participant was measured. There is no standard deviation.
  End of Trial (Week 160): number analyzed (Participants) | 21
  End of Trial (Week 160) | 3.62 (0.80)

7. Secondary Outcome: Work Limitations Questionnaire
Description: Work Limitations Questionnaire by visit. Comprised of 25 items, in 4 categories, or demands: Mental/Interpersonal, Output Tasks, Physical Tasks, and Time Management, measuring the degree to which employed individuals are experiencing limitations on-the-job due to their health problems, and health-related productivity loss. 1= All of the time (100%), 2= most of the time, 3=some of the time (about 50%), 4=slight bit of time, 5=none of the time (0%), 6=does not apply to my job. (Presenteeism). The WLQ items ask respondents to rate their level of difficulty or ability to perform specific job demands. Scale score range from 0 (limited none of the time=better outcome) to 100 (limited all of the time= worse outcome) and represent the reported amount of time in the prior two weeks respondents were limited on-the-job.
Time Frame: Baseline, Month 3, Month 6 and Every 26 weeks for up to 160 weeks
Population: All individuals for whom Work Limitations was measured. Trial was terminated early.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Elamipretide
Number analyzed (Participants) | 28
score on a scale
  Mental/Interpersonal: Baseline: number analyzed (Participants) | 12
  Mental/Interpersonal: Baseline | 67.59 (15.58)
  Mental/Interpersonal: Week 13: number analyzed (Participants) | 10
  Mental/Interpersonal: Week 13 | 71.33 (20.00)
  Mental/Interpersonal: Week 26: number analyzed (Participants) | 10
  Mental/Interpersonal: Week 26 | 72.00 (18.54)
  Mental/Interpersonal: Week 52: number analyzed (Participants) | 9
  Mental/Interpersonal: Week 52 | 75.06 (19.37)
  Mental/Interpersonal: Week 78: number analyzed (Participants) | 9
  Mental/Interpersonal: Week 78 | 70.62 (20.02)
  Mental/Interpersonal: Week 104: number analyzed (Participants) | 7
  Mental/Interpersonal: Week 104 | 68.57 (17.42)
  Mental/Interpersonal: Week 130: number analyzed (Participants) | 8
  Mental/Interpersonal: Week 130 | 66.11 (24.77)
  Mental/Interpersonal: End of Trial (Week 160): number analyzed (Participants) | 8
  Mental/Interpersonal: End of Trial (Week 160) | 74.72 (19.66)
  Output Task: Baseline: number analyzed (Participants) | 12
  Output Task: Baseline | 69.67 (20.99)
  Output Task: Week 13: number analyzed (Participants) | 10
  Output Task: Week 13 | 75.20 (21.89)
  Output Task: Week 26: number analyzed (Participants) | 10
  Output Task: Week 26 | 75.20 (18.16)
  Output Task: Week 52: number analyzed (Participants) | 9
  Output Task: Week 52 | 71.56 (18.05)
  Output Task: Week 78: number analyzed (Participants) | 8
  Output Task: Week 78 | 61.50 (20.28)
  Output Task: Week 104: number analyzed (Participants) | 6
  Output Task: Week 104 | 59.33 (25.85)
  Output Task: Week 130: number analyzed (Participants) | 8
  Output Task: Week 130 | 73.00 (22.50)
  Output Task: End of Trial (Week 160): number analyzed (Participants) | 8
  Output Task: End of Trial (Week 160) | 71.00 (19.91)
  Physical Task: Baseline: number analyzed (Participants) | 12
  Physical Task: Baseline | 56.39 (23.37)
  Physical Task Week 13: number analyzed (Participants) | 10
  Physical Task Week 13 | 58.67 (17.37)
  Physical Task Week 26: number analyzed (Participants) | 10
  Physical Task Week 26 | 55.00 (11.57)
  Physical Task Week 52: number analyzed (Participants) | 9
  Physical Task Week 52 | 52.59 (14.32)
  Physical Task Week 78: number analyzed (Participants) | 9
  Physical Task Week 78 | 57.78 (11.55)
  Physical Task Week 104: number analyzed (Participants) | 7
  Physical Task Week 104 | 56.67 (25.53)
  Physical Task Week 130: number analyzed (Participants) | 8
  Physical Task Week 130 | 58.33 (23.03)
  Physical Task: End of Trial (Week 160): number analyzed (Participants) | 8
  Physical Task: End of Trial (Week 160) | 58.75 (23.03)
  Time Management Baseline: number analyzed (Participants) | 10
  Time Management Baseline | 61.60 (23.26)
  Time Management Week 13: number analyzed (Participants) | 10
  Time Management Week 13 | 72.40 (21.54)
  Time Management Week 26: number analyzed (Participants) | 9
  Time Management Week 26 | 68.00 (24.25)
  Time Management Week 52: number analyzed (Participants) | 9
  Time Management Week 52 | 68.89 (25.83)
  Time Management Week 78: number analyzed (Participants) | 9
  Time Management Week 78 | 72.89 (21.43)
  Time Management Week 104: number analyzed (Participants) | 6
  Time Management Week 104 | 56.67 (27.76)
  Time Management Week 130: number analyzed (Participants) | 7
  Time Management Week 130 | 57.71 (29.11)
  Time Management End of Trial (Week 160): number analyzed (Participants) | 7
  Time Management End of Trial (Week 160) | 68.57 (24.92)

8. Secondary Outcome: Physician Global Assessment Score (PhGA) by Visit
Description: Physician Global Assessment- Mean Score by visit. PGA Scale asks physician to rate participant's current health status as follows: 1=Excellent, 2=Very good, 3=Good, 4=Fair, and 5=Poor. Total score ranges from 1-5. Higher score means lower health status, worse outcome; lower score means better health status, better outcome.
Time Frame: Baseline, Month 3, Month 6 and Every 26 weeks for up to 160 weeks
Population: All participants for whom PhGA was measured. Trial was terminated early.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Elamipretide
Number analyzed (Participants) | 28
score on a scale
  Baseline | 3.32 (0.61)
  Week 13: number analyzed (Participants) | 26
  Week 13 | 3.11 (0.80)
  Week 26: number analyzed (Participants) | 27
  Week 26 | 3.00 (0.73)
  Week 52: number analyzed (Participants) | 25
  Week 52 | 2.72 (0.84)
  Week 78: number analyzed (Participants) | 24
  Week 78 | 3.25 (0.79)
  Week 104: number analyzed (Participants) | 22
  Week 104 | 3.18 (0.85)
  Week 130: number analyzed (Participants) | 22
  Week 130 | 3.18 (0.73)
  Week 156: number analyzed (Participants) | 1
  Week 156 | 5.00 (NA) — Only 1 participant was measured.
  End of Study (Week 160): number analyzed (Participants) | 20
  End of Study (Week 160) | 3.40 (0.60)

9. Secondary Outcome: Physician Global Assessment (PhGA): Categorical
Description: Physician Global Assessment [PhGA] Score by Visit, Physician-reported current health status by visit. PhGA Scale is as follows: 1=Excellent, 2=Very good, 3=Good, 4=Fair, and 5=Poor. Total score ranges from 1-5. Higher score means worse health status, means worse outcome.
Time Frame: Baseline, Month 3, Month 6 and Every 26 weeks for up to 160 weeks
Population: All participants for whom PhGA was measured. Trial was terminated early.
Measure: Count of Participants; unit: Participants
Groups:
- Excellent: Number of participants the Physician rated current disease status as Excellent
- Fair: Number of participants Physician rated current disease status as Fair
- Good: Number of participants Physician rated current disease status as Good
- Poor: Number of participants Physician rated current disease status as Poor
- Very Good: Number of participants the Physician rated current disease status as Very Good
Arm/Group | Excellent | Fair | Good | Poor | Very Good
Number analyzed (Participants) | 28 | 28 | 28 | 28 | 28
Participants
  Baseline | 0 | 8 | 18 | 1 | 1
  Week 13: number analyzed (Participants) | 27 | 27 | 27 | 27 | 27
  Week 13 | 0 | 7 | 13 | 1 | 6
  Week 26: number analyzed (Participants) | 27 | 27 | 27 | 27 | 27
  Week 26 | 1 | 6 | 16 | 0 | 4
  Week 52: number analyzed (Participants) | 25 | 25 | 25 | 25 | 25
  Week 52 | 1 | 2 | 12 | 1 | 9
  Week 78: number analyzed (Participants) | 24 | 24 | 24 | 24 | 24
  Week 78 | 0 | 8 | 11 | 1 | 4
  Week 104: number analyzed (Participants) | 22 | 22 | 22 | 22 | 22
  Week 104 | 0 | 4 | 12 | 2 | 4
  Week 130: number analyzed (Participants) | 22 | 22 | 22 | 22 | 22
  Week 130 | 0 | 5 | 13 | 1 | 3
  Week 156: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1
  Week 156 | 0 | 0 | 0 | 1 | 0
  End of Study (Week 160): number analyzed (Participants) | 20 | 20 | 20 | 20 | 20
  End of Study (Week 160) | 0 | 6 | 13 | 1 | 0

10. Secondary Outcome: PMMSA Individual Items
Description: The PMMSA is a patient-reported outcome measure, assessing a participant's "worst feeling" of 10 symptoms during the last 24 hours: tiredness at rest, tiredness during activities, muscle weakness at rest, muscle weakness during activities, balance, vision, abdominal discomfort, muscle pain, numbness, and headache using a 4-point scale: 1=Not at all, 2=Mild, 3=Moderate, and 4=Severe. Max Score =40= worse outcome, Min score= 10= better outcome on scale. PMMSA Individual Items shows number or participants with mild, moderate, severe or no symptoms at all.
Time Frame: Baseline, Week 13, 26, 52, 104, 156, End of Study (Week 160)
Population: All participants for which PMMSA was measured. Trial was terminated early.
Measure: Count of Participants; unit: Participants
Arm/Group | Elamipretide
Number analyzed (Participants) | 28
Participants
  Baseline: Abdominal Discomfort: number analyzed (Participants) | 27
  Baseline: Abdominal Discomfort: Mild | 11
  Baseline: Abdominal Discomfort: Moderate | 5
  Baseline: Abdominal Discomfort: Not At All | 8
  Baseline: Abdominal Discomfort: Severe | 3
  Baseline: Balance Problems: number analyzed (Participants) | 27
  Baseline: Balance Problems: Mild | 5
  Baseline: Balance Problems: Moderate | 16
  Baseline: Balance Problems: Not At All | 1
  Baseline: Balance Problems: Severe | 5
  Baseline: Headache: number analyzed (Participants) | 27
  Baseline: Headache: Mild | 4
  Baseline: Headache: Moderate | 6
  Baseline: Headache: Not At All | 16
  Baseline: Headache: Severe | 1
  Baseline: Muscle Pain: number analyzed (Participants) | 27
  Baseline: Muscle Pain: Mild | 6
  Baseline: Muscle Pain: Moderate | 12
  Baseline: Muscle Pain: Not At All | 5
  Baseline: Muscle Pain: Severe | 4
  Baseline: Muscle Weakness at Rest: number analyzed (Participants) | 26
  Baseline: Muscle Weakness at Rest: Mild | 12
  Baseline: Muscle Weakness at Rest: Moderate | 10
  Baseline: Muscle Weakness at Rest: Not At All | 1
  Baseline: Muscle Weakness at Rest: Severe | 3
  Baseline:Muscle Weakness during Activities: number analyzed (Participants) | 27
  Baseline:Muscle Weakness during Activities: Mild | 2
  Baseline:Muscle Weakness during Activities: Moderate | 18
  Baseline:Muscle Weakness during Activities: Not At All | 0
  Baseline:Muscle Weakness during Activities: Severe | 7
  Baseline: Numbness: number analyzed (Participants) | 27
  Baseline: Numbness: Mild | 11
  Baseline: Numbness: Moderate | 2
  Baseline: Numbness: Not At All | 11
  Baseline: Numbness: Severe | 3
  Baseline: Tiredness at Rest: number analyzed (Participants) | 27
  Baseline: Tiredness at Rest: Mild | 6
  Baseline: Tiredness at Rest: Moderate | 13
  Baseline: Tiredness at Rest: Not At All | 0
  Baseline: Tiredness at Rest: Severe | 8
  Baseline: Tiredness during Activities: number analyzed (Participants) | 27
  Baseline: Tiredness during Activities: Mild | 5
  Baseline: Tiredness during Activities: Moderate | 13
  Baseline: Tiredness during Activities: Not At All | 0
  Baseline: Tiredness during Activities: Severe | 9
  Baseline: Vision Problems: number analyzed (Participants) | 27
  Baseline: Vision Problems: Mild | 8
  Baseline: Vision Problems: Moderate | 9
  Baseline: Vision Problems: Not At All | 6
  Baseline: Vision Problems: Severe | 4
  Week 13:Abdominal Discomfort: Mild | 6
  Week 13:Abdominal Discomfort: Moderate | 8
  Week 13:Abdominal Discomfort: Not At All | 11
  Week 13:Abdominal Discomfort: Severe | 3
  Week 13: Balance Problems: Mild | 11
  Week 13: Balance Problems: Moderate | 9
  Week 13: Balance Problems: Not At All | 1
  Week 13: Balance Problems: Severe | 7
  Week 13: Headache: Mild | 10
  Week 13: Headache: Moderate | 2
  Week 13: Headache: Not At All | 14
  Week 13: Headache: Severe | 2
  Week 13: Muscle Pain: Mild | 11
  Week 13: Muscle Pain: Moderate | 7
  Week 13: Muscle Pain: Not At All | 7
  Week 13: Muscle Pain: Severe | 3
  Week 13: Muscle Weakness at Rest: Mild | 13
  Week 13: Muscle Weakness at Rest: Moderate | 6
  Week 13: Muscle Weakness at Rest: Not At All | 7
  Week 13: Muscle Weakness at Rest: Severe | 2
  Week 13: Muscle Weakness during Activities: Mild | 10
  Week 13: Muscle Weakness during Activities: Moderate | 9
  Week 13: Muscle Weakness during Activities: Not At All | 3
  Week 13: Muscle Weakness during Activities: Severe | 6
  Week 13: Numbness: Mild | 6
  Week 13: Numbness: Moderate | 6
  Week 13: Numbness: Not At All | 15
  Week 13: Numbness: Severe | 1
  Week 13: Tiredness at Rest: Mild | 14
  Week 13: Tiredness at Rest: Moderate | 10
  Week 13: Tiredness at Rest: Not At All | 2
  Week 13: Tiredness at Rest: Severe | 2
  Week 13: Tiredness during Activities: Mild | 12
  Week 13: Tiredness during Activities: Moderate | 11
  Week 13: Tiredness during Activities: Not At All | 0
  Week 13: Tiredness during Activities: Severe | 5
  Week 13: Vision Problems: Mild | 11
  Week 13: Vision Problems: Moderate | 7
  Week 13: Vision Problems: Not At All | 8
  Week 13: Vision Problems: Severe | 2
  Week 26:Abdominal Discomfort: number analyzed (Participants) | 27
  Week 26:Abdominal Discomfort: Mild | 7
  Week 26:Abdominal Discomfort: Moderate | 5
  Week 26:Abdominal Discomfort: Not At All | 13
  Week 26:Abdominal Discomfort: Severe | 2
  Week 26: Balance Problems: number analyzed (Participants) | 27
  Week 26: Balance Problems: Mild | 11
  Week 26: Balance Problems: Moderate | 9
  Week 26: Balance Problems: Not At All | 1
  Week 26: Balance Problems: Severe | 6
  Week 26: Headache: number analyzed (Participants) | 27
  Week 26: Headache: Mild | 13
  Week 26: Headache: Moderate | 1
  Week 26: Headache: Not At All | 12
  Week 26: Headache: Severe | 1
  Week 26: Muscle Pain: number analyzed (Participants) | 27
  Week 26: Muscle Pain: Mild | 11
  Week 26: Muscle Pain: Moderate | 7
  Week 26: Muscle Pain: Not At All | 7
  Week 26: Muscle Pain: Severe | 2
  Week 26: Muscle Weakness at Rest: number analyzed (Participants) | 27
  Week 26: Muscle Weakness at Rest: Mild | 13
  Week 26: Muscle Weakness at Rest: Moderate | 4
  Week 26: Muscle Weakness at Rest: Not At All | 7
  Week 26: Muscle Weakness at Rest: Severe | 3
  Week 26: Muscle Weakness during Activities: number analyzed (Participants) | 27
  Week 26: Muscle Weakness during Activities: Mild | 10
  Week 26: Muscle Weakness during Activities: Moderate | 11
  Week 26: Muscle Weakness during Activities: Not At All | 1
  Week 26: Muscle Weakness during Activities: Severe | 5
  Week 26: Numbness: number analyzed (Participants) | 27
  Week 26: Numbness: Mild | 7
  Week 26: Numbness: Moderate | 3
  Week 26: Numbness: Not At All | 14
  Week 26: Numbness: Severe | 3
  Week 26: Tiredness at Rest: number analyzed (Participants) | 27
  Week 26: Tiredness at Rest: Mild | 15
  Week 26: Tiredness at Rest: Moderate | 8
  Week 26: Tiredness at Rest: Not At All | 1
  Week 26: Tiredness at Rest: Severe | 3
  Week 26: Tiredness during Activities: number analyzed (Participants) | 27
  Week 26: Tiredness during Activities: Mild | 12
  Week 26: Tiredness during Activities: Moderate | 10
  Week 26: Tiredness during Activities: Not At All | 0
  Week 26: Tiredness during Activities: Severe | 5
  Week 26: Vision Problems: number analyzed (Participants) | 27
  Week 26: Vision Problems: Mild | 6
  Week 26: Vision Problems: Moderate | 9
  Week 26: Vision Problems: Not At All | 7
  Week 26: Vision Problems: Severe | 5
  Week 52: Abdominal Discomfort: number analyzed (Participants) | 25
  Week 52: Abdominal Discomfort: Mild | 10
  Week 52: Abdominal Discomfort: Moderate | 2
  Week 52: Abdominal Discomfort: Not At All | 10
  Week 52: Abdominal Discomfort: Severe | 3
  Week 52: Balance Problems: number analyzed (Participants) | 25
  Week 52: Balance Problems: Mild | 10
  Week 52: Balance Problems: Moderate | 9
  Week 52: Balance Problems: Not At All | 1
  Week 52: Balance Problems: Severe | 5
  Week 52: Headache: number analyzed (Participants) | 25
  Week 52: Headache: Mild | 10
  Week 52: Headache: Moderate | 4
  Week 52: Headache: Not At All | 10
  Week 52: Headache: Severe | 1
  Week 52: Muscle Pain: number analyzed (Participants) | 25
  Week 52: Muscle Pain: Mild | 8
  Week 52: Muscle Pain: Moderate | 6
  Week 52: Muscle Pain: Not At All | 9
  Week 52: Muscle Pain: Severe | 2
  Week 52: Muscle Weakness at Rest: number analyzed (Participants) | 25
  Week 52: Muscle Weakness at Rest: Mild | 8
  Week 52: Muscle Weakness at Rest: Moderate | 8
  Week 52: Muscle Weakness at Rest: Not At All | 6
  Week 52: Muscle Weakness at Rest: Severe | 3
  Week 52: Muscle Weakness during Activities: number analyzed (Participants) | 25
  Week 52: Muscle Weakness during Activities: Mild | 12
  Week 52: Muscle Weakness during Activities: Moderate | 7
  Week 52: Muscle Weakness during Activities: Not At All | 1
  Week 52: Muscle Weakness during Activities: Severe | 5
  Week 52: Numbness: number analyzed (Participants) | 25
  Week 52: Numbness: Mild | 4
  Week 52: Numbness: Moderate | 5
  Week 52: Numbness: Not At All | 13
  Week 52: Numbness: Severe | 3
  Week 52:Tiredness at Rest: number analyzed (Participants) | 25
  Week 52:Tiredness at Rest: Mild | 12
  Week 52:Tiredness at Rest: Moderate | 8
  Week 52:Tiredness at Rest: Not At All | 4
  Week 52:Tiredness at Rest: Severe | 1
  Week 52:Tiredness during Activities: number analyzed (Participants) | 25
  Week 52:Tiredness during Activities: Mild | 12
  Week 52:Tiredness during Activities: Moderate | 10
  Week 52:Tiredness during Activities: Not At All | 0
  Week 52:Tiredness during Activities: Severe | 3
  Week 52:Vision Problems: number analyzed (Participants) | 25
  Week 52:Vision Problems: Mild | 8
  Week 52:Vision Problems: Moderate | 9
  Week 52:Vision Problems: Not At All | 5
  Week 52:Vision Problems: Severe | 3
  Week 78: Abdominal Discomfort: number analyzed (Participants) | 24
  Week 78: Abdominal Discomfort: Mild | 11
  Week 78: Abdominal Discomfort: Moderate | 2
  Week 78: Abdominal Discomfort: Not At All | 9
  Week 78: Abdominal Discomfort: Severe | 2
  Week 78: Balance Problems: number analyzed (Participants) | 24
  Week 78: Balance Problems: Mild | 7
  Week 78: Balance Problems: Moderate | 13
  Week 78: Balance Problems: Not At All | 1
  Week 78: Balance Problems: Severe | 3
  Week 78: Headache: number analyzed (Participants) | 24
  Week 78: Headache: Mild | 6
  Week 78: Headache: Moderate | 3
  Week 78: Headache: Not At All | 14
  Week 78: Headache: Severe | 1
  Week 78:Muscle Pain: number analyzed (Participants) | 24
  Week 78:Muscle Pain: Mild | 10
  Week 78:Muscle Pain: Moderate | 5
  Week 78:Muscle Pain: Not At All | 7
  Week 78:Muscle Pain: Severe | 2
  Week 78: Muscle Weakness at Rest: number analyzed (Participants) | 24
  Week 78: Muscle Weakness at Rest: Mild | 10
  Week 78: Muscle Weakness at Rest: Moderate | 9
  Week 78: Muscle Weakness at Rest: Not At All | 5
  Week 78: Muscle Weakness at Rest: Severe | 0
  Week 78:Muscle Weakness during Activities: number analyzed (Participants) | 24
  Week 78:Muscle Weakness during Activities: Mild | 8
  Week 78:Muscle Weakness during Activities: Moderate | 9
  Week 78:Muscle Weakness during Activities: Not At All | 2
  Week 78:Muscle Weakness during Activities: Severe | 5
  Week 78: Numbness: number analyzed (Participants) | 24
  Week 78: Numbness: Mild | 7
  Week 78: Numbness: Moderate | 3
  Week 78: Numbness: Not At All | 12
  Week 78: Numbness: Severe | 2
  Week 78:Tiredness at Rest: number analyzed (Participants) | 24
  Week 78:Tiredness at Rest: Mild | 11
  Week 78:Tiredness at Rest: Moderate | 8
  Week 78:Tiredness at Rest: Not At All | 1
  Week 78:Tiredness at Rest: Severe | 4
  Week 78:Tiredness during Activities: number analyzed (Participants) | 24
  Week 78:Tiredness during Activities: Mild | 8
  Week 78:Tiredness during Activities: Moderate | 10
  Week 78:Tiredness during Activities: Not At All | 1
  Week 78:Tiredness during Activities: Severe | 5
  Week 78: Vision Problems: number analyzed (Participants) | 24
  Week 78: Vision Problems: Mild | 10
  Week 78: Vision Problems: Moderate | 5
  Week 78: Vision Problems: Not At All | 6
  Week 78: Vision Problems: Severe | 3
  Week 104: Abdominal Discomfort: number analyzed (Participants) | 22
  Week 104: Abdominal Discomfort: Mild | 7
  Week 104: Abdominal Discomfort: Moderate | 4
  Week 104: Abdominal Discomfort: Not At All | 10
  Week 104: Abdominal Discomfort: Severe | 1
  Week 104:Balance Problems: number analyzed (Participants) | 22
  Week 104:Balance Problems: Mild | 10
  Week 104:Balance Problems: Moderate | 7
  Week 104:Balance Problems: Not At All | 1
  Week 104:Balance Problems: Severe | 4
  Week 104:Headache: number analyzed (Participants) | 22
  Week 104:Headache: Mild | 5
  Week 104:Headache: Moderate | 2
  Week 104:Headache: Not At All | 14
  Week 104:Headache: Severe | 1
  Week 104:Muscle Pain: number analyzed (Participants) | 22
  Week 104:Muscle Pain: Mild | 10
  Week 104:Muscle Pain: Moderate | 7
  Week 104:Muscle Pain: Not At All | 5
  Week 104:Muscle Pain: Severe | 0
  Week 104:Muscle Weakness at Rest: number analyzed (Participants) | 21
  Week 104:Muscle Weakness at Rest: Mild | 10
  Week 104:Muscle Weakness at Rest: Moderate | 6
  Week 104:Muscle Weakness at Rest: Not At All | 4
  Week 104:Muscle Weakness at Rest: Severe | 1
  Week 104:Muscle Weakness during Activities: number analyzed (Participants) | 22
  Week 104:Muscle Weakness during Activities: Mild | 8
  Week 104:Muscle Weakness during Activities: Moderate | 8
  Week 104:Muscle Weakness during Activities: Not At All | 3
  Week 104:Muscle Weakness during Activities: Severe | 3
  Week 104:Numbness: number analyzed (Participants) | 22
  Week 104:Numbness: Mild | 5
  Week 104:Numbness: Moderate | 2
  Week 104:Numbness: Not At All | 12
  Week 104:Numbness: Severe | 3
  Week 104: Tiredness at Rest: number analyzed (Participants) | 22
  Week 104: Tiredness at Rest: Mild | 11
  Week 104: Tiredness at Rest: Moderate | 6
  Week 104: Tiredness at Rest: Not At All | 2
  Week 104: Tiredness at Rest: Severe | 3
  Week 104:Tiredness during Activities: number analyzed (Participants) | 22
  Week 104:Tiredness during Activities: Mild | 10
  Week 104:Tiredness during Activities: Moderate | 9
  Week 104:Tiredness during Activities: Not At All | 1
  Week 104:Tiredness during Activities: Severe | 2
  Week 104: Vision Problems: number analyzed (Participants) | 22
  Week 104: Vision Problems: Mild | 7
  Week 104: Vision Problems: Moderate | 5
  Week 104: Vision Problems: Not At All | 5
  Week 104: Vision Problems: Severe | 5
  Week 130: Abdominal Discomfort: number analyzed (Participants) | 21
  Week 130: Abdominal Discomfort: Mild | 8
  Week 130: Abdominal Discomfort: Moderate | 1
  Week 130: Abdominal Discomfort: Not At All | 9
  Week 130: Abdominal Discomfort: Severe | 3
  Week 130: Balance Problems: number analyzed (Participants) | 21
  Week 130: Balance Problems: Mild | 8
  Week 130: Balance Problems: Moderate | 7
  Week 130: Balance Problems: Not At All | 1
  Week 130: Balance Problems: Severe | 5
  Week 130: Headache: number analyzed (Participants) | 21
  Week 130: Headache: Mild | 8
  Week 130: Headache: Moderate | 2
  Week 130: Headache: Not At All | 11
  Week 130: Headache: Severe | 0
  Week 130: Muscle Pain: number analyzed (Participants) | 21
  Week 130: Muscle Pain: Mild | 7
  Week 130: Muscle Pain: Moderate | 4
  Week 130: Muscle Pain: Not At All | 7
  Week 130: Muscle Pain: Severe | 3
  Week 130:Muscle Weakness at Rest: number analyzed (Participants) | 21
  Week 130:Muscle Weakness at Rest: Mild | 9
  Week 130:Muscle Weakness at Rest: Moderate | 7
  Week 130:Muscle Weakness at Rest: Not At All | 4
  Week 130:Muscle Weakness at Rest: Severe | 1
  Week 130: Muscle Weakness during Activities: number analyzed (Participants) | 21
  Week 130: Muscle Weakness during Activities: Mild | 8
  Week 130: Muscle Weakness during Activities: Moderate | 8
  Week 130: Muscle Weakness during Activities: Not At All | 1
  Week 130: Muscle Weakness during Activities: Severe | 4
  Week 130:Numbness: number analyzed (Participants) | 21
  Week 130:Numbness: Mild | 7
  Week 130:Numbness: Moderate | 3
  Week 130:Numbness: Not At All | 11
  Week 130:Numbness: Severe | 0
  Week 130:Tiredness at Rest: number analyzed (Participants) | 21
  Week 130:Tiredness at Rest: Mild | 9
  Week 130:Tiredness at Rest: Moderate | 9
  Week 130:Tiredness at Rest: Not At All | 1
  Week 130:Tiredness at Rest: Severe | 2
  Week 130: Tiredness during Activities: number analyzed (Participants) | 21
  Week 130: Tiredness during Activities: Mild | 9
  Week 130: Tiredness during Activities: Moderate | 10
  Week 130: Tiredness during Activities: Not At All | 0
  Week 130: Tiredness during Activities: Severe | 2
  Week 130:Vision Problems: number analyzed (Participants) | 21
  Week 130:Vision Problems: Mild | 7
  Week 130:Vision Problems: Moderate | 7
  Week 130:Vision Problems: Not At All | 4
  Week 130:Vision Problems: Severe | 3
  Week 156: Abdominal Discomfort: number analyzed (Participants) | 1
  Week 156: Abdominal Discomfort: Mild | 1
  Week 156: Abdominal Discomfort: Moderate | 0
  Week 156: Abdominal Discomfort: Not At All | 0
  Week 156: Abdominal Discomfort: Severe | 0
  Week 156:Balance Problems: number analyzed (Participants) | 1
  Week 156:Balance Problems: Mild | 1
  Week 156:Balance Problems: Moderate | 0
  Week 156:Balance Problems: Not At All | 0
  Week 156:Balance Problems: Severe | 0
  Week 156 Headache: number analyzed (Participants) | 1
  Week 156 Headache: Mild | 0
  Week 156 Headache: Moderate | 0
  Week 156 Headache: Not At All | 1
  Week 156 Headache: Severe | 0
  Week 156 Muscle Pain: number analyzed (Participants) | 1
  Week 156 Muscle Pain: Mild | 0
  Week 156 Muscle Pain: Moderate | 0
  Week 156 Muscle Pain: Not At All | 0
  Week 156 Muscle Pain: Severe | 1
  Week 156: Muscle Weakness at Rest: number analyzed (Participants) | 1
  Week 156: Muscle Weakness at Rest: Mild | 0
  Week 156: Muscle Weakness at Rest: Moderate | 1
  Week 156: Muscle Weakness at Rest: Not At All | 0
  Week 156: Muscle Weakness at Rest: Severe | 0
  Week 156: Muscle Weakness during Activities: number analyzed (Participants) | 1
  Week 156: Muscle Weakness during Activities: Mild | 0
  Week 156: Muscle Weakness during Activities: Moderate | 0
  Week 156: Muscle Weakness during Activities: Not At All | 0
  Week 156: Muscle Weakness during Activities: Severe | 1
  Week 156: Numbness: number analyzed (Participants) | 1
  Week 156: Numbness: Mild | 0
  Week 156: Numbness: Moderate | 1
  Week 156: Numbness: Not At All | 0
  Week 156: Numbness: Severe | 0
  Week 156:Tiredness at Rest: number analyzed (Participants) | 1
  Week 156:Tiredness at Rest: Mild | 0
  Week 156:Tiredness at Rest: Moderate | 0
  Week 156:Tiredness at Rest: Not At All | 0
  Week 156:Tiredness at Rest: Severe | 1
  Week 156:Tiredness during Activities: number analyzed (Participants) | 1
  Week 156:Tiredness during Activities: Mild | 0
  Week 156:Tiredness during Activities: Moderate | 0
  Week 156:Tiredness during Activities: Not At All | 0
  Week 156:Tiredness during Activities: Severe | 1
  Week 156:Vision Problems: number analyzed (Participants) | 1
  Week 156:Vision Problems: Mild | 0
  Week 156:Vision Problems: Moderate | 0
  Week 156:Vision Problems: Not At All | 1
  Week 156:Vision Problems: Severe | 0
  End of Study: (Week 160) Abdominal Discomfort: number analyzed (Participants) | 20
  End of Study: (Week 160) Abdominal Discomfort: Mild | 8
  End of Study: (Week 160) Abdominal Discomfort: Moderate | 2
  End of Study: (Week 160) Abdominal Discomfort: Not At All | 6
  End of Study: (Week 160) Abdominal Discomfort: Severe | 4
  End of Study: (Week 160) Balance Problems: number analyzed (Participants) | 21
  End of Study: (Week 160) Balance Problems: Mild | 9
  End of Study: (Week 160) Balance Problems: Moderate | 8
  End of Study: (Week 160) Balance Problems: Not At All | 0
  End of Study: (Week 160) Balance Problems: Severe | 4
  End of Study: (Week 160) Headache: number analyzed (Participants) | 21
  End of Study: (Week 160) Headache: Mild | 9
  End of Study: (Week 160) Headache: Moderate | 5
  End of Study: (Week 160) Headache: Not At All | 7
  End of Study: (Week 160) Headache: Severe | 0
  End of Study: (Week 160) Muscle Pain: number analyzed (Participants) | 21
  End of Study: (Week 160) Muscle Pain: Mild | 5
  End of Study: (Week 160) Muscle Pain: Moderate | 9
  End of Study: (Week 160) Muscle Pain: Not At All | 4
  End of Study: (Week 160) Muscle Pain: Severe | 3
  End of Study: (Week 160) Muscle Weakness at Rest: number analyzed (Participants) | 21
  End of Study: (Week 160) Muscle Weakness at Rest: Mild | 8
  End of Study: (Week 160) Muscle Weakness at Rest: Moderate | 7
  End of Study: (Week 160) Muscle Weakness at Rest: Not At All | 4
  End of Study: (Week 160) Muscle Weakness at Rest: Severe | 2
  End of Study: (Week 160): Muscle Weakness during Activities: number analyzed (Participants) | 21
  End of Study: (Week 160): Muscle Weakness during Activities: Mild | 3
  End of Study: (Week 160): Muscle Weakness during Activities: Moderate | 11
  End of Study: (Week 160): Muscle Weakness during Activities: Not At All | 2
  End of Study: (Week 160): Muscle Weakness during Activities: Severe | 5
  End of Study: (Week 160) Numbness: number analyzed (Participants) | 21
  End of Study: (Week 160) Numbness: Mild | 5
  End of Study: (Week 160) Numbness: Moderate | 5
  End of Study: (Week 160) Numbness: Not At All | 11
  End of Study: (Week 160) Numbness: Severe | 0
  End of Study: (Week 160) Tiredness at Rest: number analyzed (Participants) | 21
  End of Study: (Week 160) Tiredness at Rest: Mild | 7
  End of Study: (Week 160) Tiredness at Rest: Moderate | 9
  End of Study: (Week 160) Tiredness at Rest: Not At All | 1
  End of Study: (Week 160) Tiredness at Rest: Severe | 4
  End of Study: (Week 160) Tiredness during Activities: number analyzed (Participants) | 21
  End of Study: (Week 160) Tiredness during Activities: Mild | 4
  End of Study: (Week 160) Tiredness during Activities: Moderate | 10
  End of Study: (Week 160) Tiredness during Activities: Not At All | 1
  End of Study: (Week 160) Tiredness during Activities: Severe | 6
  End of Study: (Week 160): Vision Problems: number analyzed (Participants) | 21
  End of Study: (Week 160): Vision Problems: Mild | 3
  End of Study: (Week 160): Vision Problems: Moderate | 9
  End of Study: (Week 160): Vision Problems: Not At All | 6
  End of Study: (Week 160): Vision Problems: Severe | 3

11. Secondary Outcome: Total Fatigue Score_Primary Mitochondrial Myopathy Symptom Assessment (PMMSA)
Description: Change from baseline in the Total Fatigue score Primary Mitochondrial Myopathy Symptom Assessment (PMMSA) where participants report their "worst feeling" of 4 symptoms: Tiredness at rest, Tiredness during activities, Muscle weakness at rest, Muscle weakness during activities, at the end of each treatment period. Total fatigue score is sum of Q1 to Q4 only of PMMSA) and is scored as follows: 1=Not at all, 2=Mild, 3=Moderate, and 4=Severe. Total score range is 4-16; lower score means less fatigue and better outcome, higher score means more fatigue and worse outcome. Raw scores were transformed into percentages: 0-100%. Change from baseline: the lower the score, the better the outcome,=less fatigue; the higher the score, means worse outcome= more fatigue.
Time Frame: Baseline, Month 3, Month 6 and Every 26 weeks for up to 160 weeks
Population: All participants for whom PMMSA was measured. Study terminated early.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Elamipretide
Number analyzed (Participants) | 28
score on a scale
  Week 13: number analyzed (Participants) | 27
  Week 13 | -15.12 (29.33)
  Week 26: number analyzed (Participants) | 26
  Week 26 | -15.06 (29.72)
  Week 52: number analyzed (Participants) | 24
  Week 52 | -17.01 (25.36)
  Week 78: number analyzed (Participants) | 23
  Week 78 | -13.41 (31.05)
  Week 104: number analyzed (Participants) | 21
  Week 104 | -18.65 (30.15)
  Week 130: number analyzed (Participants) | 20
  Week 130 | -12.92 (31.12)
  Week 156: number analyzed (Participants) | 1
  Week 156 | 25.00 (NA) — No standard deviation because only 1 participant was measured.
  End of Trial (Week 160): number analyzed (Participants) | 20
  End of Trial (Week 160) | -8.33 (33.00)

12. Secondary Outcome: Total Fatigue Score During Activities_Primary Mitochondrial Myopathy Symptom Assessment (PMMSA)
Description: Change from baseline in the Total Fatigue during Activities score Primary Mitochondrial Myopathy Symptom Assessment (PMMSA) where participants report their "worst feeling" of 2 symptoms: Tiredness during activities, Muscle weakness during activities, at the end of each treatment period. Total fatigue score is sum of Q2 and Q4 only of PMMSA) and is scored as follows: 1=Not at all, 2=Mild, 3=Moderate, and 4=Severe. Total score range is 2-8; lower score means less fatigue and better outcome, higher score means more fatigue and worse outcome. Raw scores were transformed into percentages: 0-100%. Change from baseline: the lower the score, the better the outcome,=less fatigue; the higher the score, means worse outcome= more fatigue.
Time Frame: Baseline, Month 3, Month 6 and Every 26 weeks for up to 160 weeks
Population: All participants for whom PMMSA was measured. Study terminated early.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Elamipretide
Number analyzed (Participants) | 28
score on a scale
  Week 13: number analyzed (Participants) | 13
  Week 13 | -14.20 (29.13)
  Week 26: number analyzed (Participants) | 26
  Week 26 | -14.10 (28.55)
  Week 52: number analyzed (Participants) | 24
  Week 52 | -17.36 (25.76)
  Week 78: number analyzed (Participants) | 23
  Week 78 | -14.49 (32.30)
  Week 104: number analyzed (Participants) | 21
  Week 104 | -20.63 (28.34)
  Week 130: number analyzed (Participants) | 20
  Week 130 | -15.00 (31.94)
  Week 156: number analyzed (Participants) | 1
  Week 156 | 33.33 (NA) — Only 1 participant was measured. There is no standard deviation.
  End of Trial (Week 160): number analyzed (Participants) | 20
  End of Trial (Week 160) | -8.33 (31.30)

ADVERSE EVENTS:
Time Frame: Baseline through end of study for up to 260 weeks
Arm/Group | Elamipretide
All-Cause Mortality (participants affected / at risk) | 0/28
Serious Adverse Events (participants affected / at risk) | 8/28
Other Adverse Events (participants affected / at risk) | 28/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Elamipretide (N=28)
Pancreatitis acute (Gastrointestinal disorders) | 1
Breast cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Hemiparesis (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Cerebrovascular accident (Vascular disorders) | 1
Hereditary optic atrophy (Congenital, familial and genetic disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Ankle fracture (Injury, poisoning and procedural complications) | 1
Troponin increased (Investigations) | 1
Renal colic (Renal and urinary disorders) | 1
Urosepsis (Infections and infestations) | 1
Acute kidney injury (Renal and urinary disorders) | 1
Bacteraemia (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Bradycardia (Cardiac disorders) | 1
Intestinal obstruction (Gastrointestinal disorders) | 1
Cholelithiasis (Hepatobiliary disorders) | 1
Tibia fracture (Injury, poisoning and procedural complications) | 1
Pneumonia (Infections and infestations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Elamipretide (N=28)
Tachycardia (Cardiac disorders) | 3
Vomiting (Gastrointestinal disorders) | 5
Abdominal distension (Gastrointestinal disorders) | 3
Abdominal pain (Gastrointestinal disorders) | 3
Abdominal pain upper (Gastrointestinal disorders) | 3
Diarrhoea (Gastrointestinal disorders) | 3
Abdominal discomfort (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 2
Haemorrhoids (Gastrointestinal disorders) | 2
Impaired gastric emptying (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 2
Injection site pruritus (Gastrointestinal disorders) | 21
Injection site pruritus (General disorders) | 18
Injection site mass (General disorders) | 13
Injection site urticaria (General disorders) | 13
Injection site pain (General disorders) | 10
Injection site swelling (General disorders) | 7
Chest pain (General disorders) | 6
Fatigue (General disorders) | 6
Injection site bruising (General disorders) | 4
Injection site rash (General disorders) | 4
Pyrexia (General disorders) | 3
Chills (General disorders) | 2
Injection site haemorrhage (General disorders) | 2
Injection site induration (General disorders) | 2
Peripheral swelling (General disorders) | 2
Nasopharyngitis (Infections and infestations) | 8
Gastroenteritis viral (Infections and infestations) | 6
Urinary tract infection (Infections and infestations) | 4
Sinusitis (Infections and infestations) | 4
Upper respiratory tract infection (Infections and infestations) | 4
Influenza (Infections and infestations) | 3
Bronchitis (Infections and infestations) | 2
Ear infection (Infections and infestations) | 2
Fungal infection (Infections and infestations) | 2
Hordeolum (Infections and infestations) | 2
Pneumonia (Infections and infestations) | 2
Postoperative wound infection (Infections and infestations) | 2
Vaginal infection (Infections and infestations) | 2
Fall (Injury, poisoning and procedural complications) | 10
Concussion (Injury, poisoning and procedural complications) | 4
Contusion (Injury, poisoning and procedural complications) | 4
Ligament sprain (Infections and infestations) | 3
Skin laceration (Infections and infestations) | 3
Joint dislocation (Injury, poisoning and procedural complications) | 2
Muscle strain (Injury, poisoning and procedural complications) | 2
Thermal burn (Injury, poisoning and procedural complications) | 2
Blood lactic acid increased (Investigations) | 4
Alanine aminotransferase increased (Investigations) | 3
Eosinophil count increased (Investigations) | 3
Weight increased (Investigations) | 2
Hypokalaemia (Metabolism and nutrition disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4
Back pain (Musculoskeletal and connective tissue disorders) | 3
Muscle fatigue (Musculoskeletal and connective tissue disorders) | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2
Headache (Nervous system disorders) | 7
Dizziness (Nervous system disorders) | 3
Hypoaesthesia (Nervous system disorders) | 3
Migraine (Nervous system disorders) | 3
Neuralgia (Nervous system disorders) | 3
Dizziness postural (Nervous system disorders) | 2
Dystonia (Nervous system disorders) | 2
Syncope (Nervous system disorders) | 2
Tremor (Nervous system disorders) | 2
Anxiety (Psychiatric disorders) | 3
Depression (Psychiatric disorders) | 3
Adjustment disorder with depressed mood (Psychiatric disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 3
Apnoea (Respiratory, thoracic and mediastinal disorders) | 3
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2
Rash (Skin and subcutaneous tissue disorders) | 3
Urticaria (Skin and subcutaneous tissue disorders) | 3
Acne (Skin and subcutaneous tissue disorders) | 2
Dermal cyst (Skin and subcutaneous tissue disorders) | 2
Pruritus (Skin and subcutaneous tissue disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-29): https://cdn.clinicaltrials.gov/large-docs/38/NCT02976038/Prot_SAP_000.pdf